CLINICAL TRIAL: NCT02668341
Title: PsoBarrierEU - Barrier Analysis of Guideline-Compliant Healthcare for Psoriasis in Europe
Brief Title: Cross Sectional Analysis of Healthcare for Psoriasis in 4 European Countries
Acronym: PsoBarrier
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Sandoz (Industry)
Responsible Party: Sponsor
Other Study IDs: IVDP-405-14
Record Dates: First submitted 2015-10-12; First posted 2016-01-29 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- psoriasis patients in Denmark: non-interventional survey study in psoriasis patients in daily practice care
  Interventions: Other: non-interventional
- psoriasis patients in Spain: non-interventional survey study in psoriasis patients in daily practice care
  Interventions: Other: non-interventional
- psoriasis patients in Poland: non-interventional survey study in psoriasis patients in daily practice care
  Interventions: Other: non-interventional
- psoriasis patients in Germany: non-interventional survey study in psoriasis patients in daily practice care
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional — non-interventional survey study
  Other Names: non-interventional survey study

SUMMARY:
Analysis of barriers in psoriasis care from the patient's and the physician's perspective and generation of scientific data on the quality of health care in Denmark, Poland, Spain, and Germany

DETAILED DESCRIPTION:
Cross-sectional, non-interventional study on healthcare for psoriasis in patients and their treating physicians. Clinical data on severity as well as subjective estimates on disease burden, quality of life etc. will be collected. Data collection is planned at multiple, representative sites in fourEuropean countries with different healthcare systems with the aim to identify system-dependent and -independent barriers in guideline-compliant psoriasis care.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed psoriasis vulgaris
* age ≥ 18
* written informed consent

Exclusion Criteria:

* lack of mental, physical or linguistic ability to participate in a questionnaire survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with diagnosed psoriasis vulgaris
Sampling Method: Probability Sample
Enrollment: 1304 (Actual)
Dates: Start 2015-10; Primary Completion 2020-09 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with severe disease receiving systemic treatment | Baseline

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | Baseline
  Psoriasis disease severity, measured by validated instrument
Body Surface Area (BSA) | Baseline
  Psoriasis-affected body area, measured by physician estimate
Dermatology Life Quality Index (DLQI) | Baseline
  Quality of life assessment in dermatologic patients, measured by validated quality of life instrument
EuroQuol (EQ-5D) | Baseline
  generic quality of life assessment, measured by validated visual analogue scale
Percentage of patients with comorbidities receiving treatment. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Augustin, Prof. Dr., Study Director — Institute for Health Services Research in Dermatology and Nursing, University Medical Center Hamburg-Eppendorf, Germany
Locations (4):
- Aarhus University Hospital, Aarhus, Denmark
- Nationwide group of dermatological centers, hospitals and medical offices, Hamburg, Germany
- Medical University of Poznan, Poznan, Poland
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided